CLINICAL TRIAL: NCT03133702
Title: Characteristics of the Traumatic Forensic Cases Admitted to Emergency Department and Errors in the Forensic Reports
Brief Title: Traumatic Characteristics of the Forensic Cases Admitted to Emergency Department and Errors in the Forensic Reports
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Dr, Adiyaman University Research Hospital
Other Study IDs: ADYU 6
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Emergencies; Trauma
MeSH Terms: conditions — Emergencies; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Forensic cases — Forensic cases which were admitted to the Emergency Department

SUMMARY:
Objectives: to detect the mistakes and deficiencies of the forensic reports which was written and to detect the injury characteristics of the forensic cases applied to emergency service of a tertiary hospital.

DETAILED DESCRIPTION:
All patients who applied for reasons such as crushing, traffic accidents, firearms and explosive injuries, assault, all kinds of injuries, burns, electric shock, asphyxia, torture, child abuse, falls and other injuries, poisoning and suicide attempt are a forensic case.Traumatic forensic cases are often confronted in emergency departments, Aim to this study is to detect the mistakes and deficiencies of the forensic reports which was written and also aimed to detect the injury characteristics of the forensic cases applied to emergency department which is the most important center in region at a tertiary hospital.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic forensic cases which written a forensic report were included in study.

Exclusion Criteria:

* The forensic cases which can not be reached the forensic report and patients' emergency department chart

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatic forensic cases which applied to Emergency Department of Adıyaman University Tranining and Research Hospital, between January 01, 2014 and December 31, 2014.
Sampling Method: Non-Probability Sample
Enrollment: 4300 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Forensic cases admitted to Emergency department | one year
  Forensic cases by data obtained from medical records

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchanan A, Norko M. The forensic evaluation and report: an agenda for research. J Am Acad Psychiatry Law. 2013;41(3):359-65. PMID 24051588